CLINICAL TRIAL: NCT00250692
Title: Analgesic Effect of Nitrous Oxide in Neonates Undergoing Heel Stick
Brief Title: A Study to Test the Pain-relieving Effect of Laughing Gas in Infants
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: unknown - no record of study conduct in departmental archive
Sponsor: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 05-04-029-01
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Analgesic Affect
MeSH Terms: interventions — Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide

SUMMARY:
Our proposal is to study infants in the Neonatal Intensive Care Unit (NICU) who are undergoing a heel stick for blood sampling, a standard procedure in patient care. Currently, these infants do not get any pain relief for this procedure. Several recent clinical studies have shown the usefulness of nitrous oxide (laughing gas) for treating pain for minor procedures in children 0 to 18 years, but these effects have not been exclusively studied in the newborn and infant populations. Animal studies have questioned the anti-nociceptive (pain-blocking) effect of nitrous oxide in very young animals. It is unclear if this also applies to humans. The reason for this difference may be due to an immaturity of the neural pathways that modulate pain in the very young. The purpose of this study is to investigate whether or not nitrous oxide has an analgesic (pain-relieving) effect in infants undergoing minor procedures in the neonatal period (less than 3 months).

ELIGIBILITY:
Inclusion Criteria:

- Full-term babies up to three months old scheduled for heel stick blood draw.

Exclusion Criteria:

* preterm, difficult airway (micrognathia, cranio-facial malformation, choanal atresia, Pierre Robin syndrome, or Treacher Collins syndrome), sedated, intubated (including tracheostomy), have an oxygen requirement (FiO2>40%), anemia, bone marrow suppression, or cardiac defect

Ages: 1 Minute to 3 Months | Sex: All
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
NIPS scale
salivary cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wald, MD, Principal Investigator — UCLA Department of Anesthesiology
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States